CLINICAL TRIAL: NCT07371026
Title: The Effect of Using Distractor Cards and Thermochromic Cards on Pain, Fear, Anxiety and Procedure Time in Children Receiving Inhaler Therapy
Acronym: CALM-INH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammed Ata Nur GEÇER (Other)
Collaborators: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Muhammed Ata Nur GEÇER, MSc, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-13022260-300-1436826
Record Dates: First submitted 2026-01-05; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Acute Upper Respiratory Tract Infection; Pediatric; Pediatric Acute Respiratory Failure
Keywords: pediatrics; nebulizer therapy; thermochromic card; child; distracting card

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- thermochromic card (Experimental): The thermochromic card aims to distract the child's attention.
  Interventions: Other: thermochromic card
- distraction card (Experimental): The distraction card aims to divert the child's attention to something else.
  Interventions: Other: distraction card
- clinic's routine inhaler treatment group (No Intervention): the group in which routine inhaler therapy is applied and no additional intervention is required

INTERVENTIONS:
Other: thermochromic card — Distraction with thermochromic card
  Other Names: Termokromik kart
  Arms: thermochromic card
Other: distraction card — A distraction card is a visual aid used during medical procedures to reduce a child's perception of pain and fear by diverting their focus away from the procedure and towards the card.
  Arms: distraction card

SUMMARY:
THE EFFECT OF USİNG DİSTRACTOR CARDS AND THERMOCHROMİC CARDS ON PAİN, FEAR, ANXİETY AND PROCEDURE TİME İN CHİLDREN RECEİVİNG INHALER THERAPY.

Respiratory illnesses in children are a leading cause of childhood morbidity and mortality worldwide. Organizations such as the World Health Organization (WHO) and the Centers for Disease Control and Prevention (CDC) report that millions of children are hospitalized each year due to respiratory illnesses (He, Wang, & Zhang, 2025). A large proportion of these illnesses are caused by viral agents, and pathogens such as Respiratory Syncytial Virus (RSV), influenza, and rhinoviruses pose serious health threats to young children (Chen, Zhang, & Li, 2024).

This study will be one of the rare studies in pediatric nursing that examines the effectiveness of non-pharmacological interventions that can be applied during inhaler therapy in young age groups. The findings will contribute to nurses developing effective methods to reduce the negative emotions experienced by children during treatment. Furthermore, the first-ever use of thermochromic cards in this context in pediatric nursing will provide an innovative perspective on pediatric nursing practices.

H0: Thermochromic cards and distraction cards used during inhaler therapy have no effect on pain, fear, anxiety levels, or processing time.

Thermochromic cards used during inhaler therapy:

H1: reduce the child's pain. H2: reduce the child's fear. H3: reduce the child's anxiety level.

H4: shorten the child's processing time. Distraction cards used during inhaler therapy:

H5: reduce the child's pain. H6: reduce the child's fear. H7: reduce the child's anxiety level. H8: shorten the child's processing time.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between 4-6 years old,
* The child must be receiving inhaler treatment,
* The child must not have received IV or IM intervention before inhaler treatment,
* The child's oxygen saturation must be 95% or higher,
* The child's cognitive level and motor development must be appropriate for their age,
* The child and parents must be willing to participate in the study,
* The child and parents must be able to speak Turkish.

Exclusion Criteria:

* The child must have a cognitive or mental problem,
* The child must have special needs in terms of hearing, vision and/or speech,
* The child must have a life-threatening condition,
* The child's oxygen saturation level must be below 95%,
* The child must not be routinely receiving inhaler treatment

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Fear level before, during, and after inhalation therapy assessed by the Child Fear Scale (ÇKÖ) | Before inhalation therapy, during the procedure, and up to 5 minutes after completion of inhalation therapy
  Fear level will be assessed using the Child Fear Scale (ÇKÖ), a self-report scale consisting of six facial expressions and scored from 0 to 10 in increments of two points. Higher scores indicate greater levels of fear.
Pain intensity before, during, and after inhalation therapy assessed by the Wong-Baker FACES Pain Rating Scale | Before inhalation therapy, during the procedure, and up to 5 minutes after completion of inhalation therapy
  Pain intensity will be measured using the Wong-Baker FACES Pain Rating Scale, which consists of six facial expressions scored from 0 to 10, where higher scores represent greater pain intensity.
Anxiety level before, during, and after inhalation therapy assessed by the Child Anxiety Scale-State (ÇAS-D) | Before inhalation therapy, during the procedure, and up to 5 minutes after completion of inhalation therapy
  Anxiety level will be assessed using the Child Anxiety Scale-State (ÇAS-D), a thermometer-shaped self-report scale developed for children aged 4-10 years. Higher marked levels indicate higher state anxiety.

SECONDARY OUTCOMES:
Duration of inhalation therapy | During inhalation therapy
  Procedure duration will be recorded in minutes from the start to the completion of inhalation therapy.

IPD SHARING:
Plan to Share IPD: Undecided